CLINICAL TRIAL: NCT04634240
Title: A Randomized, Comparative Effectiveness Study of Staged Complete Revascularization With Percutaneous Coronary Intervention to Treat Coronary Artery Disease vs Medical Management Alone in Patients With Symptomatic Aortic Valve Stenosis Undergoing Elective Transfemoral Transcatheter Aortic Valve Replacement: The COMPLETE TAVR Study
Brief Title: Staged Complete Revascularization for Coronary Artery Disease vs Medical Management Alone in Patients With AS Undergoing Transcatheter Aortic Valve Replacement
Acronym: COMPLETE TAVR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, David Wood, Professor, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H20-00968
Record Dates: First submitted 2020-11-16; First posted 2020-11-18 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Aortic Stenosis; Coronary Artery Disease; Coronary Stenosis
Keywords: Transcatheter Aortic Valve Replacement; Percutaneous Coronary Intervention; Coronary Artery Disease; Aortic Stenosis
MeSH Terms: conditions — Aortic Valve Stenosis; Coronary Artery Disease; Coronary Stenosis | interventions — Percutaneous Coronary Intervention

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Complete Revascularization (Experimental): Routine PCI (percutaneous coronary intervention) of all suitable coronary artery stenoses of ≥70% in vessels ≥2.5mm in diameter.
  Interventions: Procedure: Percutaneous Coronary Intervention (PCI)
- Medical Therapy Alone (No Intervention): No revascularization of coronary artery lesions.

INTERVENTIONS:
Procedure: Percutaneous Coronary Intervention (PCI) — PCI of all qualifying lesions.
  Arms: Complete Revascularization

SUMMARY:
Patients undergoing transcatheter aortic valve replacement (TAVR) often have concomitant coronary artery disease (CAD) which may adversely affect prognosis. There is uncertainty about the benefits and the optimal timing of revascularization for such patients. There is currently clinical equipoise regarding the management of concomitant CAD in patients undergoing TAVR. Some centers perform routine revascularization with percutaneous coronary intervention (PCI) (either before or after TAVR), while others follow an alternative strategy of medical management.

The potential benefits and optimal timing of PCI in these patients are unknown. As TAVR expands to lower risk patients, and potentially becomes the preferred therapy for the majority of patients with severe aortic stenosis, the optimal management of concomitant coronary artery disease will be of increasing importance.

The COMPLETE TAVR study will determine whether, on a background of guideline-directed medical therapy, a strategy of complete revascularization involving staged PCI using drug eluting stents to treat all suitable coronary artery lesions is superior to a strategy of medical therapy alone in reducing the composite outcome of Cardiovascular Death, new Myocardial Infarction, Ischemia-driven Revascularization or Hospitalization for Unstable Angina or Heart Failure.

The study will be a randomized, multicenter, open-label trial with blinded adjudication of outcomes. Patients will be screened and consented for elective transfemoral TAVR and randomized within 96 hours of successful balloon expandable TAVR.

Complete Revascularization:

Staged PCI using third generation drug eluting stents to treat all suitable coronary artery lesions in vessels that are at least 2.5 mm in diameter and that are amenable to treatment with PCI and have a ≥70% visual angiographic diameter stenosis. Staged PCI can occur any time from 1 to 45 days post successful transfemoral TAVR.

Vs. Medical Therapy Alone:

No further revascularization of coronary artery lesions.

All patients, regardless of randomized treatment allocation, will receive guideline-directed medical therapy consisting of risk factor modification and use of evidence-based therapies. The COMPLETE TAVR study will help address the current lack of evidence in this area. It will likely impact both the global delivery of health care and the management and clinical outcomes of all patients undergoing TAVR with concomitant CAD.

ELIGIBILITY:
Inclusion Criteria:

- Symptomatic aortic valve stenosis prior to TAVR (NYHA Functional Class ≥ 2 OR Abnormal exercise test with severe SOB, abnormal BP response, or arrhythmia)

AND

- CAD defined as: at least 1 coronary artery lesion of ≥70% visual angiographic diameter stenosis in a native segment ≥2.5 mm in diameter that is not a CTO and is amenable to treatment with PCI

AND

- Consensus by the Local Multidisciplinary Heart Team that the patient is suitable for elective transfemoral TAVR with a balloon expandable transcatheter heart valve AND would receive a bypass with an anastomosis distal to the coronary artery lesion(s) if they were undergoing SAVR.

Local Multidisciplinary Heart Teams are expected to follow current clinical guidelines for selection of patients for TAVR with an eligible patient generally expected to have:

[AVA ≤ 1.0 cm2 OR AVA index ≤ 0.6 cm2/m2]

OR

[Jet velocity ≥ 4.0 m/s OR mean gradient ≥ 40 mmHg]

OR

patients without these criteria may undergo TAVR if the Local Multidisciplinary Heart Team concludes it is appropriate.

AND

- Successful transfemoral TAVR, defined as the implantation of a single transcatheter aortic valve within the past 96 hours with freedom from more than minimal aortic insufficiency, stroke, or major vascular complications.

Exclusion Criteria:

* PCI already performed within 90 days prior to TAVR or at the same time as the index transfemoral TAVR procedure
* Planned PCI of coronary artery lesion(s)
* Planned surgical revascularization of coronary artery lesion(s)
* Non-cardiovascular co-morbidity reducing life expectancy to < 5 years
* Any factor precluding 5-year follow-up
* Prior coronary artery bypass grafting surgery or surgical valve replacement
* Severe mitral regurgitation (> 3+)
* Severe left ventricular dysfunction (LVEF < 30%)
* Low coronary takeoff (high risk for coronary obstruction)
* Acute myocardial infarction within 90 days
* Stroke or transient ischemic attack within 90 days
* Renal insufficiency (eGFR < 30 ml/min) and/or renal replacement Rx
* Hemodynamic or respiratory instability

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 4000 (Estimated)
Dates: Start 2020-12-19 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Composite of Cardiovascular Death or New Myocardial Infarction or Ischemia-Driven Revascularization or Hospitalization for Unstable Angina or Heart Failure | Median follow-up of 3.5 years

SECONDARY OUTCOMES:
Cardiovascular Death or New Myocardial Infarction | Median follow-up of 3.5 years
  Deaths will be classified as cardiovascular or non-cardiovascular. All deaths with a clear cardiovascular or unknown cause, will be classified as cardiovascular. However, within cardiovascular deaths, hemorrhagic deaths will be clearly identified. Only deaths due to a documented non-cardiovascular cause (e.g., cancer) will be classified as non-cardiovascular.
  Myocardial Infarction will be defined according to the 4th Universal Definition of Myocardial Infarction, with modification for Type 4a (PCI-related) and Type 5 (CABG-related) as defined for the ISCHEMIA trial and as used in the COMPLETE trial.
Transaortic gradient immediately post-TAVR (echocardiographically-derived vs. direct invasive measurement) | Immediately post-TAVR
Transaortic Gradient Reclassification | Median follow-up of 3.5 years
  Proportion of patients developing echocardiographic aortic gradient ≥20 mmHg who are found to have a gradient < 20 mmHg on direct hemodynamic assessment.
VARC-3 Hemodynamic Valve Deterioration Reclassification | Median follow-up of 3.5 years
  Proportion of patients developing ≥ moderate echocardiographic VARC-3 valve deterioration reclassified to < moderate VARC-3 valve deterioration using direct invasive methods, including mean gradient and valve area.
Severe Patient Prosthesis Mismatch (PPM) Reclassification | Median follow-up of 3.5 years
  Proportion of patients with echocardiographic severe PPM immediately post-TAVR, reclassified as non-severe PPM using direct invasive methods.
Composite of CV Death, New MI, IDR or Hospitalization for UA or for HF in patients with PPM and elevated gradients vs those without | Median follow-up of 3.5 years
  Deaths: will be classified as cardiovascular or non-cardiovascular. All deaths with a clear cardiovascular or unknown cause, will be classified as cardiovascular. However, within cardiovascular deaths, hemorrhagic deaths will be clearly identified. Only deaths due to a documented non-cardiovascular cause (e.g., cancer) will be classified as non-cardiovascular.
  Myocardial Infarction: will be defined according to the 4th Universal Definition of Myocardial Infarction, with modification for Type 4a (PCI-related) and Type 5 (CABG-related) as defined for the ISCHEMIA trial and as used in the COMPLETE trial.
  Hospital admission: for protocol-defined unstable angina, new/worsening NYHA Class IV heart failure, or for protocol-defined Ischemia-driven revascularization, among patients with patient prosthesis mismatch (PPM), elevated echocardiography-derived transaortic gradients and elevated direct invasive transaortic gradient vs those without.
Composite outcome of mean echocardiographic gradient ≥ 20mmHg, severe PPM, ≥ moderate AR, thrombosis, endocarditis, and aortic valve re-intervention | Median follow-up of 3.5 years
Cardiovascular Death | Median follow-up of 3.5 years
New Myocardial Infarction | Median follow-up of 3.5 years
Ischemia-Driven Revascularization | Median follow-up of 3.5 years
Hospitalization for Unstable Angina or Heart Failure | Median follow-up of 3.5 years
All-cause Mortality | Median follow-up of 3.5 years
  Includes deaths from both cardiac and non-cardiac causes
Stroke | Median follow-up of 3.5 years
  Defined as the presence of a new focal neurologic deficit thought to be vascular in origin, with signs or symptoms lasting more than 24 hours. It is strongly recommended (but not required) that an imaging procedure such as CT scan or MRI be performed. Stroke will be further classified as ischemic, hemorrhagic or type uncertain.
Bleeding | Median follow-up of 3.5 years
  Clinically overt, symptomatic bleeding with at least one of the following criteria:
  * Fatal, or
  * Symptomatic intracranial hemorrhage, or
  * Retroperitoneal hemorrhage, or
  * Intraocular hemorrhage leading to significant vision loss, or
  * Decrease in hemoglobin of 3.0 g/dL (with each blood transfusion unit counting for 1.0 g/dL of Hb) or requiring transfusion of two or more units of red blood cells or equivalent of whole blood.
  * Requiring surgical intervention to stop the bleeding
Angina status | Median follow-up of 3.5 years
  As evaluated by the Seattle Angina Questionnaire
Economic evaluation | Median follow-up of 3.5 years
  Includes health resource utilization, costs, and cost-effectiveness
Patient-reported outcomes | Median follow-up of 3.5 years
  Health-related quality of life as evaluated by the Kansas City Cardiomyopathy Questionnaire at baseline, 30 days, 6 months, 1 year, and annually thereafter.
Contrast-associated acute kidney injury | Median follow-up of 3.5 years
  An absolute rise in serum creatinine of greater than or equal to 44 μmol/L from baseline and/or a relative rise in serum creatinine of ≥25% compared to baseline at any time between 48hrs and 96hrs post-procedure.
Fluoroscopic time for Staged PCI procedure | During PCI procedure
  Total time under fluoroscopy
Contrast Utilization for Stages PCI Procedure | During PCI procedure

CONTACTS AND LOCATIONS:
Overall Officials: David A Wood, MD, Principal Investigator — CCI-CIC, University of British Columbia
Locations (72):
- United States (55):
  - Huntsville Heart Center, Huntsville, Alabama
  - Arizona Cardiovascular Research, Phoenix, Arizona
  - Veteran Affairs Palo Alto Health Care System, Palo Alto, California
  - Loma Linda University, Redlands, California
  - Santa Barbara Cottage Hospital, Santa Barbara, California
  - Torrance Memorial Medical Center, Torrance, California
  - JFK Medical Center, Atlantis, Florida
  - Baptist Health Jacksonville, Jacksonville, Florida
  - Miami Cardiac and Vascular/Baptist Hospital, Miami, Florida
  - Piedmont, Atlanta, Georgia
  - Northeast Georgia Health System, Gainesville, Georgia
  - St. Alphonsus Regional Medical Center, Boise, Idaho
  - Ascension Alexian Brothers, Chicago, Illinois
  - Midwest Cardiovascular Research and Education Foundation, Elkhart, Indiana
  - Parkview Research Center, Fort Wayne, Indiana
  - University of Kansas Medical Center, Kansas City, Kansas
  - Midwest Heart and Vascular, Overland Park, Kansas
  - Cardiovascular Research Institute of Kansas, Wichita, Kansas
  - Tufts Medical, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - Sparrow Clinical Research Institute, Lansing, Michigan
  - William Beaumont Hospital, Royal Oak, Michigan
  - Ascension St. Mary's, Saginaw, Michigan
  - St. Joseph Mercy Health System, Ypsilanti, Michigan
  - University of Minnesota Medical Center, Minneapolis, Minnesota
  - CentraCare Heart and Vascular Center, Saint Cloud, Minnesota
  - Boone Hospital, Columbia, Missouri
  - St. Louis University, St Louis, Missouri
  - Missouri Baptist, St Louis, Missouri
  - Bryan Heart, Lincoln, Nebraska
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Our Lady of Lourdes, Camden, New Jersey
  - Valley Hospital, Ridgewood, New Jersey
  - University at Buffalo, Buffalo, New York
  - NYU Langone Hospital - Long Island, Mineola, New York
  - Mount Sinai, New York, New York
  - Columbia University Medical Center, New York, New York
  - St. Joseph's Hospital, Syracuse, New York
  - Montefiore Medical Center, The Bronx, New York
  - Novant Health Heart and Vascular Institute, Charlotte, North Carolina
  - Summa Health System, Akron, Ohio
  - Mount Carmel, Columbus, Ohio
  - Oklahoma Heart, Oklahoma City, Oklahoma
  - Kaiser Permanente Northwest, Clackamas, Oregon
  - Rhode Island Hospital, Providence, Rhode Island
  - Methodist Le Bonheur Healthcare, Germantown, Tennessee
  - Ballad Health CVA Heart Institute, Kingsport, Tennessee
  - Parkwest Medical Center, Knoxville, Tennessee
  - Cardiovascular Surgery Clinic/Baptist Memorial, Memphis, Tennessee
  - HCA Houston Healthcare Medical Center, Houston, Texas
  - Baylor Scott & White Plano, Plano, Texas
  - Baylor Scott & White Round Rock, Round Rock, Texas
  - University of Vermont Medical Center, Burlington, Vermont
  - Bellin Health System, Green Bay, Wisconsin
  - Ascension Columbia St. Mary's, Milwaukee, Wisconsin
- Canada (17):
  - University of Alberta, Mazankowski Heart Institute, Edmonton, Alberta
  - Royal Columbian Hospital, New Westminster, British Columbia
  - Vancouver General Hospital, Vancouver, British Columbia
  - Centre for Cardiovascular Innovation-Centre d'Innovation Cardiovasculaire (CCI-CIC), Vancouver, British Columbia
  - St. Paul's Hospital, Vancouver, British Columbia
  - Saint Boniface, Winnipeg, Manitoba
  - New Brunswick Heart, Saint John, New Brunswick
  - Queen Elizabeth II Health Sciences Centre, Halifax, Nova Scotia
  - Hamilton Health Sciences, Hamilton, Ontario
  - Ottawa Heart, Ottawa, Ontario
  - Sunnybrook Hospital, Toronto, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - Montréal Heart, Montreal, Quebec
  - Centre Hospitalier de l'Université de Montréal, Montreal, Quebec
  - Sacré-Coeur, Montreal, Quebec
  - CIUSSS de l'Estrie-CHUS, Sherbrooke, Quebec
  - Prairie Vascular, Regina, Saskatchewan

IPD SHARING:
Plan to Share IPD: No